CLINICAL TRIAL: NCT03687827
Title: A Randomised, Cross-over, Open-label, Multi-centre Trial Comparing the Effect of Insulin Degludec and Insulin Glargine 100U/mL, With or Without OADs in Subjects With Type 2 Diabetes Using Flash Glucose Monitoring
Brief Title: A Research Study to Compare the Effect of Insulin Degludec and Insulin Glargine on Blood Sugar Levels in People With Type 2 Diabetes - the SWITCH PRO Study
Acronym: SWITCH PRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-4419; U1111-1203-0580 (Other: World Health Organization (WHO)); 2017-004047-20 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin degludec (Experimental): Participants will receive insulin degludec in period 1 and 2 in a cross-over manner.
  Interventions: Drug: Insulin degludec
- Insulin glargine (Active Comparator): Participants will receive insulin glargine in period 1 and 2 in a cross-over manner.
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin degludec — Participants will receive insulin degludec U100 subcutaneous (s.c.) injection once daily for 36 weeks. Doses will be adjusted according to the fasting self-measured plasma glucose (SMPG) values. Participants earlier treated with one or more allowed oral antidiabetic drug(s) (OAD(s)), should continue their pre-trial OAD(s) treatment throughout the trial.
  Other Names: Tresiba®
  Arms: Insulin degludec
Drug: Insulin glargine — Participants will receive insulin glargine U100 s.c. injection once daily for 36 weeks. Doses will be adjusted according to the fasting SMPG values. Participants earlier treated with one or more allowed OAD(s), should continue their pre-trial OAD(s) treatment throughout the trial.
  Other Names: Lantus®
  Arms: Insulin glargine

SUMMARY:
This study compares the effect on blood sugar levels of two medicines: insulin degludec and insulin glargine in people with type 2 diabetes. Participants will be treated with insulin degludec and insulin glargine during two different periods. Which treatment participants get first is decided by chance. Both medicines are approved for use in humans and available on the market. They can already be prescribed by participants' doctors. Participants will get pre-filled insulin pens to inject these insulins with. The study will last for about 41 weeks. Participants will visit the clinic 13 times and have 27 phone calls with the study doctor or study staff. At 12 of the clinic visits they will take blood samples. In order to evaluate the changes in participants' blood sugar level over time, participants will be asked to wear a small (35 millimetres (mm) x 5 mm) sensor on the back of participants' upper arm 3 times during the study. Each time participants must wear the sensor for 2 weeks. This sensor is called FreeStyle Libre Pro®. It has a very small tip which is 0.4 mm thick and is inserted 5 mm under participants' skin. Please note that participants will not be able to see the sensor readings while wearing it. The study doctor will show participants the readings when participants return to the clinic. Participants will be asked to fill in a diary in between visits. Participants will have contact with the study doctor or study staff each week. This is to adjust the dose of participants' study medicines and to ensure that participants are well. Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus greater than or equal to 180 days prior to the day of screening
* Subjects fulfilling at least one of the below criteria:
* Experienced at least one severe hypoglycaemic episode within the last year prior to screening (according to the American Diabetes Association definition, January 2018)*
* Moderate renal impairment defined as estimated glomerular filtration rate value of 30-59 mL/min/1.73 m^2 as defined by Kidney Disease Improving Global Outcomes 2012 at screening
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8 at screening
* Treated with insulin for more than 5 years
* Episode of hypoglycaemia (defined a glucose alert value of 70 mg/dL (3.9 mmol/L) or less, i.e., Level 1) within the last 12 weeks prior to screening visit
* Treated with any basal insulin greater than or equal to 90 days prior to the day of screening with or without any of the following anti-diabetic drugs:
* Metformin
* Dipeptidyl peptidase-4 inhibitor
* Sodium-glucose co-transporter 2 inhibitor
* Alpha-glucosidase-inhibitors (acarbose)
* Thiazolidinediones
* Marketed oral combination products only including the products listed above
* HbA1c less than or equal to 9.5% (80 mmol/mol) at screening confirmed by central laboratory analysis
* Body mass index less than or equal to 45 kg/m^2 *Hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, intermittent bolus insulin treatment for periods of no longer than 14 days are permitted prior to the day of screening
* Anticipated initiation or change in concomitant medications known to affect weight or glucose metabolism (e.g., treatment with orlistat, thyroid hormones, or corticosteroids)
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (60):
- United States (31):
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Hamden, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Kalispell, Montana
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Dakota Dunes, South Dakota
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Kerrville, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
- Canada (9):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Markham, Ontario
  - Novo Nordisk Investigational Site, Oakville, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Warsaw
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Slovakia (9):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Bytča
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Malacky
  - Novo Nordisk Investigational Site, Nové Mesto nad Váhom
  - Novo Nordisk Investigational Site, Nové Zámky
  - Novo Nordisk Investigational Site, Trebišov
  - Novo Nordisk Investigational Site, Trnava
  - Novo Nordisk Investigational Site, Žilina
- South Africa (6):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Derived] Goldenberg RM, Aroda VR, Billings LK, Donatsky AM, Frederiksen M, Klonoff DC, Kalyanam B, Bergenstal RM. Correlation Between Time in Range and HbA1c in People with Type 2 Diabetes on Basal Insulin: Post Hoc Analysis of the SWITCH PRO Study. Diabetes Ther. 2023 May;14(5):915-924. doi: 10.1007/s13300-023-01389-2. Epub 2023 Mar 11. PMID 36905485
- [Derived] Goldenberg RM, Aroda VR, Billings LK, Christiansen ASL, Meller Donatsky A, Parvaresh Rizi E, Podgorski G, Raslova K, Klonoff DC, Bergenstal RM. Effect of insulin degludec versus insulin glargine U100 on time in range: SWITCH PRO, a crossover study of basal insulin-treated adults with type 2 diabetes and risk factors for hypoglycaemia. Diabetes Obes Metab. 2021 Nov;23(11):2572-2581. doi: 10.1111/dom.14504. Epub 2021 Aug 16. PMID 34322967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 5 countries as follows:
  Canada: 10 sites, Poland: 5 sites, Slovakia: 10 sites, South Africa: 7 sites, United States of America: 34 sites
Pre-assignment Details: This was a cross-over trial. The trial included a 2-week run-in period (which was after the screening visit) for eligibility assessment in regard to adherence to FGM requirements. The participants were randomized into one of two treatment sequences.
Groups:
- Sequence A: Insulin Degludec 100U/mL Then Insulin Glargine 100U/mL: Participants were to receive a subcutaneous (s.c.) injection of Insulin degludec 100U/mL (Units per milliliter) once daily (in treatment period 1), followed by a s.c. injection of Insulin glargine 100U/mL once daily (in treatment period 2) with or without oral anti-diabetic drugs using flash glucose monitoring. Each treatment period consisted of a 16-week titration period followed by a 2-week maintenance period.
- Sequence B: Insulin Glargine 100U/mL Then Insulin Degludec 100U/mL: Participants were to receive a subcutaneous (s.c.) injection of Insulin glargine 100U/mL once daily (in treatment period 1), followed by a s.c. injection of Insulin degludec 100U/mL once daily (in treatment period 2) with or without oral anti-diabetic drugs using flash glucose monitoring. Each treatment period consisted of a 16-week titration period followed by a 2-week maintenance period.
Period: Treatment Period 1
Arm/Group | Sequence A: Insulin Degludec 100U/mL Then Insulin Glargine 100U/mL | Sequence B: Insulin Glargine 100U/mL Then Insulin Degludec 100U/mL
Started | 249 | 249
Full Analysis Set (FAS) | 249 | 249
Safety Analysis Set (SAS) | 249 | 249
Per Protocol Set | 219 | 229
Completed | 235 | 241
Not Completed | 14 | 8
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 7 | 3
Period: Treatment Period 2
Arm/Group | Sequence A: Insulin Degludec 100U/mL Then Insulin Glargine 100U/mL | Sequence B: Insulin Glargine 100U/mL Then Insulin Degludec 100U/mL
Started | 235 | 241
Completed | 230 | 238
Not Completed | 5 | 3
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Overall Study: Participants were to receive subcutaneous (s.c.) injection of Insulin degludec 100U/mL once daily followed by a s.c. injection of Insulin glargine 100U/mL once daily in 2 treatment periods with or without oral anti-diabetic drugs using flash glucose monitoring. Each treatment period consisted of a 16-week titration period followed by a 2-week maintenance period.
Arm/Group | Overall Study
Number analyzed (Participants) | 498
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259
  Male | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100
  Not Hispanic or Latino | 398
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 23
  Black or African American | 39
  White | 415
  Other | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent in Glycaemic Target Range 70-180 mg/dL (3.9-10.0 mmol/L) Both Inclusive, Using Flash Glucose Monitoring (FGM)
Description: The percentage of time spent in glycaemic target range was calculated as the number of recorded measurements in glycaemic target range (70-180 milligrams per deciliter [mg/dL] (3.9-10.0 millimoles per litre [mmol/L]), both inclusive) divided by the total number of recorded measurements. The endpoint is based on data recorded by FGM system. It was required that at least 70% of the planned FGM measurements during weeks 16-17 and weeks 34-35 were available for endpoint data to be included in the analysis.
Time Frame: During the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2)
Population: Per protocol (PP) analysis set - The PP analysis set consisted of subjects that stayed on assigned treatment until and completed FGM assessment at visits 21 and 39 respectively.
  Complete FGM assessment was specified as subjects having at least 70% of 2 weeks FGM measurements per maintenance period (2 * 960 measurements).
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Groups:
- Insulin Degludec 100U/mL: Participants were to receive a subcutaneous (s.c.) injection of insulin degludec 100U/mL, once daily, in any of the treatment period, with or without oral anti-diabetic drugs using flash glucose monitoring. Each treatment period consisted of a 16-week titration period followed by a 2-week maintenance period.
- Insulin Glargine 100U/mL: Participants were to receive a subcutaneous (s.c.) injection of insulin glargine 100U/mL, once daily, in any of the treatment period, with or without oral anti-diabetic drugs using flash glucose monitoring. Each treatment period consisted of a 16-week titration period followed by a 2-week maintenance period.
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
Percentage of Time | 72.11 (0.74) | 70.68 (0.74)
Statistical Analysis 1: Comparison: Insulin Degludec 100U/mL vs Insulin Glargine 100U/mL; Test type: Superiority — Superiority is confirmed if non-inferiority is confirmed and the lower limit of the two-sided 95% confidence interval is entirely above zero; p = 0.0321, t-test, 2 sided; Estimated treatment difference = 1.43, 95% CI 2-sided [0.12 to 2.74]
Statistical Analysis 2: Comparison: Insulin Degludec 100U/mL vs Insulin Glargine 100U/mL; Test type: Non-Inferiority — A non-inferiority margin of -0.83% has been applied, corresponding to 0.2 hours/24 hours; Estimated treatment difference = 1.43, 95% CI 2-sided [0.12 to 2.74]

2. Secondary Outcome: Time Spent in Tight Glycaemic Target Range 70-140 mg/dL (3.9-7.8 mmol/L) Both Inclusive, Using Flash Glucose Monitoring
Description: The percentage of time spent in tight glycaemic target range 70-140 mg/dL (3.9-7.8 mmol/L) both inclusive, during the 2-week maintenance periods using FGM (visit 9-21 (week 16-17) and visit 37-39 (week 34-35)).
Time Frame: During the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2).
Population: Per protocol (PP) analysis set - The PP analysis set consisted of subjects that stayed on assigned treatment until and completed FGM assessment at visits 21 and 39 respectively.
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
Percentage of Time | 52.97 (0.82) | 51.45 (0.82)

3. Secondary Outcome: Time Spent in Nocturnal Glycaemic Target Range 70-140 mg/dL (3.9-7.8 mmol/L) Both Inclusive, in the Nocturnal Period (00:01 am - 05:59 am Both Inclusive) Using Flash Glucose Monitoring
Description: Percentage of time spent in nocturnal glycaemic target range 70-140 mg/dL (3.9-7.8 mmol/L) both inclusive, in the nocturnal period (00:01 am - 05:59 am both inclusive) during the 2-week maintenance periods using FGM (visit 19-21 (week 16-17) and visit 37-39 (week 34-35)).
Time Frame: During the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of Time
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
Percentage of Time | 15.15 (0.26) | 14.91 (0.26)

4. Secondary Outcome: Level of Glycated Haemoglobin (HbA1c) - Percentage
Description: Level of HbA1c after two weeks of maintenance periods (Visit 19-21 (week 16-17) and Visit 37-39 (week 34-35)).
Time Frame: After the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycated haemoglobin
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
Percentage of glycated haemoglobin | 7.10 (0.04) | 7.16 (0.04)

5. Secondary Outcome: Level of Glycated Haemoglobin (HbA1c) - mmol/Mol
Description: Level of HbA1c after two weeks of maintenance periods (Visit 19-21 (week 16-17) and Visit 37-39 (week 34-35)).
Time Frame: After the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimoles per mole (mmol/mol)
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
millimoles per mole (mmol/mol) | 54.10 (0.42) | 54.78 (0.42)

6. Secondary Outcome: Mean Glucose Levels Using Flash Glucose Monitoring (FGM)
Description: Mean glucose levels (mmol/L) during the 2-week maintenance periods using FGM (visit 19-21 (week 16-17) and visit 37-39 (week 34-35)).
Time Frame: During the 2-week maintenance period: weeks 16-17 (period-1) and weeks 34-35 (period-2).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
Number analyzed (Participants) | 448 | 448
mmol/L | 7.57 (0.08) | 7.61 (0.08)

ADVERSE EVENTS:
Time Frame: From the randomization (week 0) up to end of treatment (week 36) and follow up (week 37).
Description: Safety Analysis Set was defined as all participants that were randomized and treated with at least one dose of trial drug after randomization.
Arm/Group | Insulin Degludec 100U/mL | Insulin Glargine 100U/mL
All-Cause Mortality (participants affected / at risk) | 0/490 | 1/484
Serious Adverse Events (participants affected / at risk) | 26/490 | 23/484
Other Adverse Events (participants affected / at risk) | 0/490 | 0/484
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec 100U/mL (N=490) | Insulin Glargine 100U/mL (N=484)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (3)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Scan myocardial perfusion abnormal (Investigations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03687827/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03687827/SAP_001.pdf